CLINICAL TRIAL: NCT06204380
Title: An Observational Study on the Identification of Prescription Patterns of STAFEN Cap., Changes in Blood Lipid Concentration, and Statin-related Muscle Symptoms in Korean Patients With Mixed Dyslipidemia
Brief Title: An Observational Study on the Identification of Prescription Patterns of STAFEN Cap
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-STAF-401
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study on the identification of prescription patterns of STAFEN Cap., changes in blood lipid concentration, and statin-related muscle symptoms in Korean patients with mixed dyslipidemia

DETAILED DESCRIPTION:
This study aims to observe the effectiveness of STAFEN capsule such as changes in blood lipid concentration and safety including statin-related muscle symptoms, and prescription patterns under daily clinical treatment in patients who have been prescribed STAFEN capsules for the treatment of complex dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. A patient diagnosed with mixed dyslipidemia
3. A patient who was first prescribed a STAFEN cap. for the purpose of treating mixed dyslipidemia according to the clinician's judgment
4. A patient who voluntarily agreed in writing to this study

Exclusion Criteria:

1. Pregnant women, lactating women, or those planning to conceive
2. A person who is prohibited from administering the STAFEN cap. under the permit
3. If the person in charge of other clinical studies and the person in charge deems it inappropriate to be the subject of this clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Prescribed STAFEN Cap. for the Treatment of Mixed Dyslipidemia
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Target triglyceride rate at 6 months of STAFEN capsule prescription compared to baseline | at 6 months of STAFEN capsule prescription compared to baseline
  Target triglyceride rate at 6 months of STAFEN capsule prescription compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Heebaek Park, Principal Investigator — delphoe clinic
Locations (1):
- Delphoe Clinic, Gangneung-si, South Korea